CLINICAL TRIAL: NCT05902598
Title: Phase 3 Study to Evaluate the Efficacy and Safety of ARO-APOC3 in Chinese Adults With Familial Chylomicronemia Syndrome
Brief Title: A Phase 3 Study of VSA001 in Chinese Adults With Familial Chylomicronemia Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSA001-3001
Record Dates: First submitted 2023-05-31; First posted 2023-06-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-03

CONDITIONS: Familial Chylomicronemia Syndrome
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- VSA001 25 mg (Experimental): VSA001 25 mg every 3 months
  Interventions: Drug: VSA001 injection
- VSA001 25 mg matching placebo (Placebo Comparator): VSA001 25 mg matching placebo，every 3 months
  Interventions: Drug: Placebo
- VSA001 50 mg (Experimental): VSA001 50 mg every 3 months
  Interventions: Drug: VSA001 injection
- VSA001 50 mg matching placebo (Placebo Comparator): VSA001 50 mg matching placebo，every 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSA001 injection — also referred to as ARO-APOC3
  Other Names: ARO-APOC3
  Arms: VSA001 25 mg; VSA001 50 mg
Drug: Placebo — Matching VSA001 injection
  Other Names: Normal saline
  Arms: VSA001 25 mg matching placebo; VSA001 50 mg matching placebo

SUMMARY:
This is a randomized, double-blinded, placebo controlled, two periods phase 3 clinical study. The primary objective of the study is to evaluate the efficacy and safety of VSA001 injection in Chinese adults with familial chylomicronemia syndrome (FCS). A total of approximately 30 participants will be enrolled in the study.

DETAILED DESCRIPTION:
Familial chylomicronemia syndrome (FCS) is a severe and ultrarare genetic disease, with a prevalence of approximately 1 in 1,000,000, often caused by various monogenic mutations. FCS leads to extremely high fasting triglyceride (TG) levels, typically over 900 mg/dL. Such severe elevations lead to various serious signs and symptoms including acute pancreatitis (which can be fatal), chronic daily abdominal pain, type 2 diabetes mellitus, hepatic steatosis, and cognitive issues.

APOC3 is an 8.8 kilodalton (kDa) protein component of triglyceride-rich lipoproteins (TRLs) such as very-low-density lipoprotein cholesterol (VLDL-C), intermediate density lipoprotein cholesterol (IDL-C), chylomicrons, high-density lipoprotein cholesterol (HDL-C), and remnant particle lipoproteins. APOC3 is synthesized predominantly in hepatocytes. It inhibits the hydrolysis of TG on TRLs at the muscle and adipose tissue capillary level through inhibition of lipoprotein lipase (LPL), and delays clearance of lipoprotein remnants by the liver by inhibiting hepatocyte receptor-mediated uptake. APOC3 functions as a key regulator of fasting and postprandial plasma TG levels.

VSA001 is a synthetic, double-stranded, hepatocyte-targeted RNA interference (RNAi) trigger (also referred to as a small interfering RNA [siRNA]) designed to specifically silence messenger RNA (mRNA) transcripts from the APOC3 gene using an RNAi mechanism. Given the important role of APOC3 in serum TG level modulation and its primary source of synthesis in hepatocytes, reduction of APOC3 through a hepatocyte-targeted RNAi strategy is likely to reduce circulating TG, benefiting several patient populations, including patients with FCS.

ELIGIBILITY:
Inclusion Criteria:

* Males or nonpregnant (who do not plan to become pregnant), nonlactating females ≥18 years of age
* Able and willing to provide written informed consent prior to the performance of any study-specific procedures
* Fasting TG ≥10 mmol/L (~880 mg/dL) at screening, that is refractory to standard lipid lowering therapy (sample drawn after at least the minimum time on stable lipid-lowering regimen described in protocol). Two repeat tests are allowed to qualify.
* A diagnosis of FCS based on a documented history of fasting TG levels in excess of 1000 mg/dL on repeated testing (for at least one prior occasions), and at least one of the following:

  1. A supportive genetic test (from a source-verifiable medical record or based on screening genotype). Supportive genetic testing includes but is not limited to homozygous, compound heterozygous, or double heterozygote for loss-of-function or otherwise inactivating mutations in genes affecting lipoprotein lipase activity including LPL, APOC2, APOA5, GPIHBP1, GPD1, or LMF1; or evidence of low LPL activity (<20% of normal) based on source-verifiable documentation; or
  2. Documented history of recurrent episodes of acute pancreatitis, not caused by alcohol or cholelithiasis; or
  3. Documented history of recurrent hospitalizations for severe abdominal pain without other explainable cause; or
  4. Documented history of childhood pancreatitis; or
  5. Family history of hypertriglyceridemia-induced pancreatitis
* Willing to follow dietary counseling as per PI judgment based on local standard of care, consistent with an intake of ≤20 g of fat per day during the study
* If on medications for management of type 2 diabetes, or other medications specified in protocol, the dosing regimen must be stable before collection of qualifying lipid parameter at screening.
* Participants with a medical history of clinical atherosclerotic cardiovascular disease (ASCVD) or those with elevated 10-year ASCVD risk (eg, ≥7.5% per American Heart Association / American College of Cardiology risk calculator) must be on appropriate lipid-lowering therapy as per local standard of care (ie, including moderate to high intensity statin, as indicated) prior to collection of qualifying TG levels.
* Participants of childbearing potential must agree to use a highly effective form of contraception in addition to a male condom, during the study and for at least 24 weeks after the last dose of IP. Women of childbearing potential on a hormonal contraceptive must be stable on the medication for ≥2 menstrual cycles prior to Day 1. Men must not donate sperm during the study and for at least 24 weeks after the last dose of IP.

Exclusion Criteria:

* Current use or use within the last 365 days from Day 1 of any hepatocyte-targeted siRNA or antisense oligonucleotide molecule
* Diabetes mellitus with any of the following:
* Newly diagnosed within 12 weeks of screening
* HbA1c ≥9.0% at screening
* Active pancreatitis within 12 weeks before Day 1
* History of acute coronary syndrome event within 24 weeks of Day 1
* History of major surgery within 12 weeks of Day 1
* Any of the following laboratory values at screening:

  1. ALT or AST ≥3×ULN at screening
  2. Total bilirubin ≥1.5×ULN (if the participant has a prior diagnosis and documentation of Gilbert's syndrome, then total bilirubin must be ≤3 mg/dL at screening)
  3. Estimated glomerular filtration rate <30 mL/min/1.73 m2 at screening, using the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) creatinine equation
  4. Spot urine protein/spot urine creatinine ratio greater than 3 grams per day
  5. Clinically significant abnormality in prothrombin time, partial thromboplastin time, or INR
* Uncontrolled hypertension (blood pressure >160/100 mmHg at screening); if untreated, participant may be rescreened once hypertension is treated and controlled
* Use of any of the following:

  1. Systemic use of corticosteroids or anabolic steroids within 4 weeks prior to Day 1 or planned use during the study
  2. GLP-1 receptor agonists
  3. Plasma apheresis within 4 weeks prior to Day 1 or planned during the study
  4. Blood donation of 50 to 499 mL within 4 weeks of collection of qualifying lipid parameter collection or of >499 mL within 8 weeks of qualifying lipid parameter collection
* On treatment with HIV antiretroviral therapy (Note: determination of HIV status is not a required study procedure)
* Seropositive (hepatitis B surface antigen [HBsAg] +) for hepatitis B virus (HBV) or hepatitis C virus (HCV) (HCV seropositivity requires positive test for antibodies confirmed with positive test for HCV RNA)
* New York Heart Association (NYHA) Class III or IV heart failure or last known ejection fraction of <30%
* Clinical evidence of primary hypothyroidism (screening TSH > ULN and free T4<LLN), primary subclinical hypothyroidism (screening TSH > ULN and free T4 WNL), or secondary hypothyroidism (screening TSH < LLN and free T4< LLN)
* History of hemorrhagic stroke within 24 weeks of first dose
* History of bleeding diathesis or coagulopathy
* Current diagnosis of nephrotic syndrome
* Unwilling to limit alcohol consumption to within moderate limits for the duration of the study, as follows: not more than 14 units per week for women and men (1 unit approximately corresponds to 80 mL of wine, 200 mL of beer, or 25 mL of 40% alcohol)
* History of malignancy within the last 2 years prior to the date of consent requiring systemic treatment except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer. Currently receiving systemic cancer treatment(s) or, in the PI's opinion, at risk of relapse for recent cancer.
* Use of an investigational agent or device within 30 days or within 5 half-lives, based on plasma PK (whichever is longer) prior to Day 1 or current participation in an interventional investigational study. Participants previously exposed to ARO-APOC3 or ARO-ANG3 will require a washout period of at least 1 year from last dose.
* Any concomitant medical or psychiatric condition or social situation or any other situation that, in the PI's judgment, would make it difficult to comply with protocol requirements or put the participant at additional safety risk.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of Fasting Triglyceride (TG) by Month 10 | Baseline, month 10
  Percent change from baseline at Month 10 in fasting TG

SECONDARY OUTCOMES:
Change of Fasting TG at Months 10 and 12 (Averaged) | Baseline, Months 10 and 12 (averaged)
  Percent change from baseline at Months 10 and 12 (averaged) in fasting TG
Change of Fasting APOC3 by Month 10 | Baseline, month 10
  Percent change from baseline at Month 10 in fasting APOC3
Change of Fasting APOC3 by Month 12 | Baseline, month 12
  Percent change from baseline at Month 12 in fasting serum APOC3
Change of Fasting Serum Non-high Density Lipoprotein Cholesterol (Non-HDL-C) and HDL-C by Month 10 | Baseline, month 10
  Percent change from baseline at Month 10 in fasting serum non-high density lipoprotein cholesterol (non-HDL-C) and HDL-C
Change of Fasting Serum TG, Non-HDL-C, and HDL-C by Month 12 | Baseline, Month 12
  Percent change from baseline at Month 12 in fasting serum TG, non-HDL-C, and HDL-C
Participants Achieving Fasting Serum TG of <500 mg/dL at Month 10 | Month 10
  Proportion of participants achieving fasting serum TG of <500 mg/dL at Month 10
Participants Achieving Fasting Serum TG of <500 mg/dL at Month 12 | Month 12
  Proportion of participants achieving fasting serum TG of <500 mg/dL at Month 12
Change From Baseline at Each Scheduled Assessment in Fasting Serum TG up to Month 12 | From baseline up to Month 12
  Change from baseline at each scheduled assessment in fasting serum TG up to Month 12(including month 1,2,3,4,5,6,7,8,9,10,11,12)
Percent Change From Baseline at Each Scheduled Assessment in Fasting Serum TG up to Month 12 | From baseline up to Month 12
  Percent change from baseline at each scheduled assessment in fasting serum TG up to Month 12(including month 1,2,3,4,5,6,7,8,9,10,11,12)
Incidence of TEAEs in the Participants | From treatment with VSA001 to 12 months
  Incidence of TEAEs in the participants
Incidence of Positively Adjudicated Events of Acute Pancreatitis | From treatment with VSA001 to 12 months
  Any AEs and SAEs reported by the investigator during the study that were consistent with acute pancreatitis events were adjudicated by the blinded Data Safety Committee based on the Atlanta Classification for Acute Pancreatitis 2013 for fulfillment of any 2 of the following 3 criteria:
  1. Abdominal pain consistent with symptoms of acute pancreatitis (acute episodes of persistent, severe upper abdominal pain often radiating to the back)
  2. Serum lipase activity (or amylase activity) ≥3 × upper limit of normal (ULN)
  3. Characteristic findings of acute pancreatitis on contrast-enhanced computed tomography (CECT) or magnetic resonance imaging (MRI) or transabdominal ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Dong YOU, MD., PhD., Study Chair — Visirna Therapeutics HK Limited
Locations (1):
- Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No